CLINICAL TRIAL: NCT06984627
Title: An Open-label Phase 2 Study to Investigate the Efficacy and Safety of Rilzabrutinib in Adult Participants With Graves' Disease
Brief Title: A Study to Investigate the Efficacy and Safety of Rilzabrutinib in Adult Participants With Graves' Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY18663; 2025-521023-75 (Registry Identifier: CTIS); U1111-1316-0208 (Other Grant/Funding Number: ICTRP)
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Graves' Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rilzabrutinib dose 1 (Experimental): Rilzabrutinib
  Interventions: Drug: Rilzabrutinib dose 1
- Rilzabrutinib dose 2 (Experimental): Rilzabrutinib
  Interventions: Drug: Rilzabrutinib dose 2

INTERVENTIONS:
Drug: Rilzabrutinib dose 1 — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: SAR444671
  Arms: Rilzabrutinib dose 1
Drug: Rilzabrutinib dose 2 — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: SAR444671
  Arms: Rilzabrutinib dose 2

SUMMARY:
This is a parallel group, Phase 2, 2-arm study to measure the treatment effect and safety of rilzabrutinib dose 1 or rilzabrutinib dose 2 in participants with Graves' disease, with and without Graves' orbitopathy, aged 18 years or older.

Study details include:

* Screening period (up to 4 weeks).
* Treatment period (up to 16 weeks).
* Follow-up period (4 weeks). The number of visits will be up to 13.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a confirmed diagnosis of Graves' disease with active hyperthyroidism, with or without active Graves' orbitopathy at the time of screening.
* A subset of participants will have a diagnosis of active Graves' orbitopathy, as confirmed by ophthalmic exam at screening and a clinical activity score (CAS) ≥3 for the most severely affected eye, and associated with one or more of the following: lid retraction ≥2 mm, moderate or severe soft tissue involvement, proptosis ≥2 mm, and/or intermittent or constant diplopia.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* History of hyperthyroidism not caused by Graves' disease (eg, hyperthyroidism due to toxic multinodular goiter, autonomous thyroid nodule, acute inflammatory thyroiditis).
* History of thyroid storm or at high risk of developing thyroid storm as determined by evaluating clinician.
* Enlarged thyroid goiter causing upper airway obstruction and/or requiring surgical intervention during the study period.
* For participant with Graves' orbitopathy, requires immediate surgical ophthalmological intervention or is planning corrective surgery/irradiation during the course of the study.
* Sight threatening Graves' orbitopathy or decreased visual acuity due to optic neuropathy within the last 6 months.
* Corneal decompensation unresponsive to medical management.
* Onset of Graves' orbitopathy symptoms >9 months prior to baseline. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in FT4 levels | At Week16
  Free thyroxine

SECONDARY OUTCOMES:
Percent change from baseline in FT3 levels | At Week16
  Free triiodothyronine
Proportion of participants with FT4 levels within normal limits | At Week16
Proportion of participants with FT3 levels within normal limits | At Week16
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs) and withdrawals due to TEAEs during the study period | Up to week 20

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (3):
  - Investigational Site Number : 1240003, Calgary, Alberta
  - Investigational Site Number : 1240002, Surrey, British Columbia
  - Investigational Site Number : 1240001, Sherbrooke, Quebec
- Germany (2):
  - Investigational Site Number : 2760002, Essen
  - Investigational Site Number : 2760001, Frankfurt
- Italy (3):
  - Investigational Site Number : 3800001, Milan, Milano
  - Investigational Site Number : 3800003, Palermo
  - Investigational Site Number : 3800002, Pisa
- Spain (2):
  - Investigational Site Number : 7240002, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240001, Pamplona, Navarre
- United Kingdom (2):
  - Investigational Site Number : 8260003, Milton Keynes, Buckinghamshire
  - Investigational Site Number : 8260001, Newcastle upon Tyne, England

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PDY18663 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26684&tenant=MT_SNY_9011